CLINICAL TRIAL: NCT07239739
Title: Effect of Triple Antibiotic Paste and Calcium Hydroxide on the Rate of Healing of Periapical Lesions in Single-Rooted Teeth: A Randomized Controlled Trial
Brief Title: Comparing Two Medicines for Healing Jaw Bone Infections After Root Canal Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faiz ur rahman (Other)
Responsible Party: Sponsor-Investigator, Faiz ur rahman, Postgraduate Resident, Department of Operative Dentistry, College of Physicians and Surgeons Pakistan
Organization: College of Physicians and Surgeons Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCD-Endo-001
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Periapical Lesion; Periapical Periodontitis
Keywords: Triple Antibiotic Paste,; Calcium Hydroxide,; Periapical Healing; Intracanal Medicament
MeSH Terms: conditions — Periapical Periodontitis | interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple Antibiotic Paste (TAP) (Experimental): TAP placed as intracanal medicament following chemo-mechanical preparation; temporary restoration maintained for several weeks
  Interventions: Drug: Triple Antibiotic Paste; Drug: Calcium Hydroxide (Ca(OH)2)
- Calcium Hydroxide Group (Active Comparator): Calcium Hydroxide intracanal dressing placed following chemo-mechanical preparation; sealed temporarily
  Interventions: Drug: Triple Antibiotic Paste; Drug: Calcium Hydroxide (Ca(OH)2)

INTERVENTIONS:
Drug: Triple Antibiotic Paste — Intracanal medicament paste composed of Ciprofloxacin, Metronidazole, and Minocycline. Placed in the root canal for several weeks.
Drug: Calcium Hydroxide (Ca(OH)2) — Standard intracanal medicament with high pH, used for its antibacterial and tissue-stimulating properties. Placed in the root canal for several weeks

SUMMARY:
This study compares two commonly used intracanal medicaments-Triple Antibiotic Paste and Calcium Hydroxide-in patients with infected single-rooted teeth. The purpose is to determine which medicament promotes faster healing of periapical lesions after root canal treatment by measuring reduction in lesion size and improvement in bone density over 3, 6, and 12 months.

DETAILED DESCRIPTION:
This single-center, parallel-arm, randomized controlled trial aims to directly compare the efficacy of Triple Antibiotic Paste (TAP) and Calcium Hydroxide (CH) as intracanal medicaments on the rate of healing of periapical lesions in single-rooted teeth. Systemically healthy adults (18-65 years) with a diagnosis of pulpal necrosis and asymptomatic apical periodontitis or chronic apical abscess, presenting with a radiographically evident periapical radiolucency (≥2mm), will be enrolled. Following informed consent, chemomechanical preparation, and randomization, participants will receive either TAP (Ciprofloxacin:Metronidazole:Minocycline) or CH as the intracanal medicament. The primary outcome is the rate of healing, quantified by the percentage reduction in periapical lesion area and improvement in bone density scores assessed on standardized periapical radiographs or CBCT scans at 3, 6, and 12-month follow-ups. Secondary outcomes include clinical resolution (absence of pain, tenderness, sinus tract) and radiographic resolution (restoration of normal periapical architecture). Data will be analyzed using intention-to-treat analysis, with repeated-measures ANOVA to compare healing trajectories between groups.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy adult patients between 18 and 65 years of age.

Presence of a single-rooted tooth diagnosed with pulpal necrosis and asymptomatic apical periodontitis or chronic apical abscess.

Radiographic evidence of a distinct periapical radiolucency with a minimum diameter of 2mm.

The involved tooth must be deemed restorable after endodontic treatment.

Patient willingness and ability to provide informed consent and comply with the follow-up schedule

Exclusion Criteria:

Patients under 18 or over 65 years of age.

Presence of systemic diseases known to affect bone metabolism or immune response (e.g., uncontrolled diabetes).

Pregnancy or lactation.

Known allergies to any components of Triple Antibiotic Paste or calcium hydroxide.

Teeth with previous root canal treatment, internal/external root resorption, root fractures, or non-endodontic periapical pathology.Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in Periapical Lesion Area | Baseline, 3 months, 6 months, 12 months
  Percentage reduction in the area (mm²) of the periapical radiolucency from baseline, as measured on standardized periapical radiographs or CBCT scans.

SECONDARY OUTCOMES:
Change in Periapical Bone Density Score | Baseline, 3 months, 6 months, 12 months
  Improvement in a standardized bone density score or grayscale value of the periapical bone from baseline

IPD SHARING:
Plan to Share IPD: No